CLINICAL TRIAL: NCT01265745
Title: A Phase I, Double-blind, Randomized, Placebo Controlled, Dose Escalation Study of Valortim® (MDX-1303) Administered Intravenously (IV) as a 120 Minute Infusion in Healthy, Normal Subjects
Brief Title: Dose Escalation Study of Valortim® (MDX-1303) Administered Intravenously (IV) in Healthy, Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAthene, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 0036-10-01; HHSN272200700033C (Other: HHSN); BAA-NIH-NIAID-DMID-07-37 (Other Grant/Funding Number: BAA-NIH-NIAID-DMID-07-37)
Record Dates: First submitted 2010-12-17; First posted 2010-12-23 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Anthrax
Keywords: Phase I
MeSH Terms: conditions — Anthrax | interventions — Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valortim (Active Comparator): Valortim 1mg,5mg,10mg
  Interventions: Biological: MDX1303
- Placebo (Placebo Comparator): Saline solution will be used as the placebo
  Interventions: Drug: Normal Saline for Injection

INTERVENTIONS:
Drug: Normal Saline for Injection — Equivalent amounts to subjects weight, once over 120 minutes
  Arms: Placebo
Biological: MDX1303 — a sterile solution at a protein concentration of 25 mg/mL: 20 mM sodium citrate, 50 mM sodium chloride, 3.0% mannitol, 50 µM diethylenetriamine pentacetic acid and 0.06% polysorbate 80 at pH 6.5. A tubular, clear glass vial, filled with a 5 mL dose of colorless to pale yellow solution. The vial is sealed with a 20 mm stopper and white flip-off seal.
  Arms: Valortim

SUMMARY:
Valortim is the name of the experimental drug that volunteers will receive in this study. Valortim may also be called MDX-1303. Experimental means that the drug is not yet approved by the Food and Drug Administration (FDA). Valortim is a monoclonal antibody (laboratory-made immune system molecule) for the treatment of inhalation anthrax (when the infection starts in the lungs). Valortim works by attaching itself to part of the anthrax toxin preventing the toxin from doing damage to cells. This study is being conducted to see if Valortim given over 120 minutes is safe and tolerable. This study will take place in five parts: Screening Phase, Check-in Phase (the day you arrive at Quintiles to start the study), Treatment Phase (the time when you receive the study medication), Follow-up Phase (the time after you receive the study medication) and Final Visit.

DETAILED DESCRIPTION:
Twenty-eight subjects will be recruited and entered into one of three dose groups 1mg/kg, 5mg/kg, 10mg/kg or placebo. Subjects will be stagger dosed into one of the three groups and randomly assigned to receive Valortim or saline. Subjects will reside in the clinical trial Phase I Unit from Day -1 through Day 2. After discharge on Day 2, all subjects will return to the Phase I unit 7 times at specified time points over an additional 130 days post-dosing (133 days total participation from check-in on Day -1)or placebo.

ELIGIBILITY:
Inclusion Criteria:

1.Subject must have read, understood, and provided written informed consent 2.Subjects should be in generally good health, based upon pre-study medical history, physical examination, laboratory testing and ECG 3.Laboratory screening values (i.e., hematology, clinical chemistries and urinalysis tests) must be within study-defined ranges 4.No detectable antibody to B. anthracis Protective Antigen (PA-IgG) as measured by ELISA testing at study Screening 5.Women of childbearing potential and sexually active males may be enrolled if protocol specific contraceptives or practices are met 6.Agreement to not receive any vaccinations Day -1 through to 29 days post dosing. Vaccination against B. anthracis is prohibited during the study.8.Body Mass Index (BMI) ≥ 19 and ≤ 30. 9. Abstinence from alcohol for 24 hours prior to study drug

Exclusion Criteria:

1. Prior known or suspected exposure to B. anthracis 2. Prior vaccination for B. anthracis 3.Prior exposure to Valortim as part of a previous clinical trial 4.Immunoglobulin E (IgE) level at screening that is above the upper limit of normal per the laboratory's reference range 5. History of drug or alcohol abuse, i.e., having been treated either in an in-patient or out-patient facility within 12 months of study Screening 6. Outward signs of active allergies or upper respiratory infection 7. History of dizziness or fainting upon standing (orthostatic hypotension) which, in the opinion of the Investigator, may interfere with safety evaluations 8. Positive drug result and/or positive alcohol result at time of study Screening or at Day -1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety | 133 days
  * Determination of changes from baseline for clinical laboratory tests and urinalysis, body temperature, heart rate, blood pressure, respiratory rate, physical examination and electrocardiogram (ECG).
  * Occurrence and evaluation of adverse events and serious adverse events.

SECONDARY OUTCOMES:
Pharmacokinetics | 133 days
  Evaluation of the pharmacokinetics/pharmacodynamics of Valortim in healthy human volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Schutz, MD, Principal Investigator — Quintiles Phase I Services; Valeire D Riddle, MD, Study Director — Sponsor Medical Monitor
Locations (1):
- Quintiles Phase I Unit, Overland Park, Kansas, United States